CLINICAL TRIAL: NCT02841098
Title: " Endarterectomy Combined With Optimal Medical Therapy Versus Optimal Medical Therapy Alone in Patients With Asymptomatic Severe Atherosclerotic Carotid Artery Stenosis at Higher-than-average Risk of Ipsilateral Stroke "
Brief Title: " Endarterectomy Combined With Optimal Medical Therapy (OMT) vs OMT Alone in Patients With Asymptomatic Severe Atherosclerotic Carotid Artery Stenosis at Higher-than-average Risk of Ipsilateral Stroke "
Acronym: ACTRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Hôpitaux Universitaires Paris Ile-de-Franc Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D15-P010
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Asymptomatic Carotid Artery Stenosis
Keywords: Carotid stenosis,stroke,endarterectomy,medical therapy
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotid endarterectomy combined with optimal medical therapy (Experimental): Carotid endarterectomy (CEA) combined with optimal medical therapy (OMT)
  Interventions: Other: Carotid endarterectomy (CEA) combined with optimal medical therapy (OMT)
- Optimal medical therapy (OMT) (Active Comparator): Optimal medical therapy (OMT)
  Interventions: Drug: Optimal medical therapy alone

INTERVENTIONS:
Other: Carotid endarterectomy (CEA) combined with optimal medical therapy (OMT) — Carotid endarterectomy (CEA) combined with optimal medical therapy (OMT) (Surgery and Drug)
  Arms: Carotid endarterectomy combined with optimal medical therapy
Drug: Optimal medical therapy alone — Optimal medical therapy alone
  Arms: Optimal medical therapy (OMT)

SUMMARY:
The purpose of this study is to determine whether carotid surgery combined with optimal medical therapy improves long-term survival free of ipsilateral stroke in patients with asymptomatic carotid stenosis at higher-than-average risk of ipsilateral stroke when compared with optimal medical therapy alone.

DETAILED DESCRIPTION:
Carotid artery stenosis >= 50% affects about 3% of subjects >= 60 years and accounts for up to 15% of all ischemic strokes. Overall, patients with asymptomatic carotid stenosis have a low risk of ipsilateral stroke on modern medical therapy. It is therefore uncertain whether the benefit of carotid surgery still justifies the perioperative risk of stroke or death, and whether revascularisation is good value for money considering competing demands on health services. Several imaging techniques have been developed to identify patients with asymptomatic carotid stenosis at higher-than-average risk of ipsilateral stroke. Specifically, the presence of transcranial Doppler (TCD)-detected embolic signals, intraplaque haemorrhage on magnetic resonance imaging, TCD-measured impaired cerebral vasomotor reserve or rapid stenosis progression have all been shown to involve an at least 3-fold higher risk of ipsilateral stroke. However, before recommendations for clinical practice can be made regarding the use of these tools, their utility must be demonstrated in a formal randomised clinical trial. Our hypothesis is that the use of these predictors can identify a subset of patients with asymptomatic carotid stenosis who could benefit from prophylactic endarterectomy.

Carotid endarterectomy The procedure will be carried out with the technique routinely used by each surgeon. Operative reports and perioperative complications will be collected. CEA will have to be performed as soon as possible, within 60 days after randomization.

Optimal medical therapy OMT will be applied to all patients and started immediately after randomisation.

OMT will be defined by the adhoc committee and follow relevant guidelines. It will include:

* Antiplatelet therapy. If the patient requires anticoagulation for any reason (e.g. atrial fibrillation), the patient should be treated with an appropriate anticoagulant according to the practice at the centre as an alternative to antiplatelet therapy.
* Antihypertensive treatment, if required, to achieve a target blood pressure < 140/90 mmHg (higher targets may be defined by the OMT committee for selected conditions, e.g. contralateral carotid occlusion) Application of structured programs, such as stepped-care approach using ranking of antihypertensive drugs will be used.
* High-dose statin treatment (target LDL < 0.7 g/l). A stepped-care approach with raking of lipid-lowering drugs will also be used.
* Patients smoking at the time of randomisation will be encouraged to stop and join a smoking cessation and support program.
* Other lifestyle modification: reduction of alcohol consumption, choosing healthy food, increasing regular physical activity, reduction of body weight if relevant.

OMT may be modified during the course of the trial to take account revised guidelines or new evidence.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or over
* No ipsilateral stroke or TIA within 180 days of randomization
* Atherosclerotic carotid stenosis between 70 and 99% (NASCET method)
* At least one of the following markers of ipsilateral stroke risk:

  * Silent brain infarction on MRI, DWi, consistent with embolism from or hemodynamic consequences of the qualifyiing stenosis
  * History of contralateral TIA or ischemic stroke due to atherosclerotic carotid disease
  * Predominantly echolucent plaque on ultrasound
  * Rapid (within 1 year) carotid stenosis progresion
  * TCD-detected microembolic signals
  * Impairment of TCD-measured cerebral vasomotor reserve
  * Intraplaque haemorrhage on magnetic resonance imaging
  * Rapid and severe stenosis progression
* Patient is able and willing to give informed consent

Exclusion Criteria:

* Previous revascularization procedure in the artery to be randomised
* Patients not suitable for endarterectomy due to anatomical factors
* Carotid stenosis caused by non-atherosclerotic disease e.g. neck radiotherapy or fibromuscular disease
* Patients who have had contralateral carotid artery or vertebral artery or intracranial artery revascularisation within 6 weeks prior to randomisation
* Patients with planned revascularisation of the contralateral carotid artery or a vertebral artery or an intracranial artery within 6 weeks after randomisation or the date of CEA
* Patients who have had coronary artery bypass grafting within 3 months prior to randomisation or other major surgery within 6 weeks prior to randomisation
* Patients with planned coronary artery bypass grafting or other major surgery within 6 weeks after CEA of the artery considered for treatment in the trial
* Patients with pre-existing disability (modified Rankin score greater than 2)
* Patients who have a low 5-year life expectancy (see appendix for definition)
* Patients intolerant or allergic to all of the medications available for OMT
* Patients in clinical trials of investigational medicinal products or who have been in clinical trials within the last 4 months will not be enrolled unless otherwise agreed
* Patients who are known to be pregnant
* Patients unwilling or unable to participate in follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Ipsilateral stroke or procedural stroke or death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any ipsilateral stroke within 6 years after randomization or procedural (within 30 days after revascularization) stroke or death

SECONDARY OUTCOMES:
Any stroke or procedural death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any stroke within 6 years after randomization or procedural death (within 30 days after revascularization)
Any disabling or fatal stroke or procedural death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any disabling or fatal stroke within 6 years after randomization or procedural death (within 30 days after revascularization)
Any stroke or TIA or procedural death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any stroke or TIA within 6 years after randomization or procedural death within 6 years after randomization
Any stroke or death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any stroke or death within 6 years after randomization
Myocardial infarction | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Myocardial infarction within 6 years after randomization
Any death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any death within 6 years after randomization
Cardiovascular death | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Cardiovascular death within 6 years after randomization
Any hospitalisation for vascular disease | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Any hospitalisation for vascular disease within 6 years after randomization
Cranial nerve palsy attributed to revascularisation | M1
  Cranial nerve palsy attributed to revascularisation within 30 days after revascularization
Haematoma caused by treatment requiring surgery, transfusion or prolonging hospital stay | M1
  Haematoma caused by treatment requiring surgery, transfusion or prolonging hospital stay within 30 days after revascularization
Further revascularisation of the randomised artery after the initial attempt. | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Further revascularisation of the randomised artery after the initial attempt.
Carotid revascularisation | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Carotid revascularisation during follow-up other than that allocated at randomisation
New cerebral infarction or haemorrhage | M24
  New cerebral infarction or haemorrhage on MRI at 2 years
Increase in white-matter changes | M0, M24
  Increase in white-matter changes on MRI at 2 years.
Cognitive impairment | M0, M24
  Cognitive impairment assessed by the Montreal Cognitive Assessment (MoCA) with adjustment for demographic factors.
Depression | M0, M24
  Depression measured by the Centre for Epidemiologic Studies Depression (CES-D) Scale.
Health-related quality of life | M0, M24
  Health-related quality of life measured using the European Quality Of Life (EQ-5D).
Disability | M0, M24
  Disability measured by the modified Rankin scale with structured interview
Achievement of goals for each of the components of optimal medical treatment | M1, M6, M12, M18, M24, M30, M36, M42, M48, M54, M60, M66, M72
  Achievement of goals for each of the components of optimal medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis MAS, Study Director — CHSA
Locations (23):
- France (23):
  - Centre Hospitalier régional de Besançon, Hôpital Jean Minjoz, Besançon
  - CHU Bordeaux, Groupe Hospitalier Pellegrin, Bordeaux
  - CHRU La Cavale Blanche, Brest
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHU Dijon-Bourgogne, Dijon
  - CHU de Grenoble, Grenoble
  - Hôpital Mignot - CH Versailles, Le Chesnay
  - CHRU de Lille, Lille
  - Hôpital Neurologique Pierre Wertheimer GHE, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nice, Hôpital Pasteur 2, Nice
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Antoine, Paris
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Centre Hospitalier Sainte-Anne, Paris
  - Centre Hospitalier Bichat-Claude Bernard, Paris
  - CHU La Milétrie, Poitiers
  - Hôpital Pontchaillou CHU Rennes, Rennes
  - CHU de Rouen, Hôpital Charles Nicolle, Rouen
  - Hôpital Nord CHU Saint-Etienne, Saint-Etienne
  - CHU de Strasbourg, Hôpital de Hautpierre, Strasbourg
  - CHU de Toulouse Hôpital Pierre-Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided